CLINICAL TRIAL: NCT03658265
Title: Effect of Exercise Training at Different Timeline on Shoulder Dysfunction in Patients After Breast Cancer Modified Radical Mastectomy: A Randomized Controlled Trial
Brief Title: Effects of Exercise Training at Different Timeline on Shoulder Dysfunction After Breast Cancer Modified Radical Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wuhan University (Other)
Responsible Party: Principal Investigator, Qing Shu, Principal Investigator, Wuhan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRE2018013
Record Dates: First submitted 2018-08-29; First posted 2018-09-05 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Shoulder Dysfunction; Breast Cancer; Modified Radical Mastectomy
Keywords: breast cancer modified radical mastectomy; shoulder dysfunction; Rehabilitation Training
MeSH Terms: conditions — Breast Neoplasms | interventions — Lead

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 7 days SIE plus 4 weeks PRE (Active Comparator): Participants in this group will start shoulder isotonic exercise 7 days after surgery and begin progressive resistance exercise 4 weeks after surgery.
  Interventions: Other: 7 days SIE plus 4 weeks PRE
- 7 days SIE plus 3 weeks PRE (Experimental): Participants in this group will start shoulder isotonic exercise 7 days after surgery and begin progressive resistance exercise 3 weeks after surgery.
  Interventions: Other: 7 days SIE plus 3 weeks PRE
- 3 days SIE plus 4 weeks PRE (Experimental): Participants in this group will start shoulder isotonic exercise 3 days after surgery and begin progressive resistance exercise 4 weeks after surgery.
  Interventions: Other: 3 days SIE plus 4 weeks PRE
- 3 days SIE plus 3 weeks PRE (Experimental): Participants in this group will start shoulder isotonic exercise 3 days after surgery and begin progressive resistance exercise 3 weeks after surgery.
  Interventions: Other: 3 days SIE plus 3 weeks PRE

INTERVENTIONS:
Other: 7 days SIE plus 4 weeks PRE — Shoulder isotonic exercise (SIE)：exercise methods for shortening and relaxing the muscles around the shoulder joint.
  Progressive resistance exercise (PRE)：A training method that gradually increases the resistance, which will increase the muscle capacity.
  Arms: 7 days SIE plus 4 weeks PRE
Other: 7 days SIE plus 3 weeks PRE — Shoulder isotonic exercise (SIE)：exercise methods for shortening and relaxing the muscles around the shoulder joint.
  Progressive resistance exercise (PRE)：A training method that gradually increases the resistance, which will increase the muscle capacity.
  Arms: 7 days SIE plus 3 weeks PRE
Other: 3 days SIE plus 4 weeks PRE — Shoulder isotonic exercise (SIE)：exercise methods for shortening and relaxing the muscles around the shoulder joint.
  Progressive resistance exercise (PRE)：A training method that gradually increases the resistance, which will increase the muscle capacity.
  Arms: 3 days SIE plus 4 weeks PRE
Other: 3 days SIE plus 3 weeks PRE — Shoulder isotonic exercise (SIE)：exercise methods for shortening and relaxing the muscles around the shoulder joint.
  Progressive resistance exercise (PRE)：A training method that gradually increases the resistance, which will increase the muscle capacity.
  Arms: 3 days SIE plus 3 weeks PRE

SUMMARY:
Patients who underwent modified radical mastectomy were enrolled in the study. 200 subjects were randomly divided into 4 groups: 7 days postoperative shoulder isotonic training + 4 weeks postoperative progressive resistance training group, postoperative 7 Isometric training for the shoulder joint + progressive resistance training for 3 weeks after surgery group, 3 days postoperative isotope training + 4 weeks postoperative progressive resistance training group, 3 days postoperative shoulder isotonic training + postoperative 3 Weekly progressive resistance training group. The effects of interventional rehabilitation at different time points on the recovery of shoulder function after breast cancer operation were observed. The results of the study will provide evidence-based evidence for the time point of intervention in early functional exercise after modified radical mastectomy for breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 25 and 75 years;
2. Diagnosed with breast cancer by pathological diagnosis, the time of diagnosis and the time of inclusion are less than 6 weeks;
3. Patients undergoing modified radical mastectomy: mastectomy includes unilateral total breast or breast-conserving surgery, as well as dissection of the affected axillary lymph nodes, but does not include sentinel lymph node biopsy;
4. Postoperative chemotherapy or radiation therapy according to the condition;
5. No other malignant tumors within 5 years;
6. No physical therapy related contraindications;
7. Signing informed consent.

Exclusion Criteria:

1. The result of SLNB is negative who did not receive ALND;
2. Received breast reconstruction surgery (prosthesis, latissimus dorsi, etc.);
3. Combined tumor metastasis with other tissues and organs (liver, kidney, lung, brain, etc.);
4. Combined severe heart disease, cerebrovascular disease, and mental illness;
5. Patients with shoulder joint dysfunction before surgery;
6. Unable to understand the rehabilitation training program provided by doctors or physiotherapists.

Ages: 25 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 200 (Actual)
Dates: Start 2018-09-10 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Constant-Murley Shoulder Score | 1 weeks after surgery
  The shoulder function was evaluated by the total score of the Constant-Murley Shoulder Score Questionnaire, which ranged from 0 to 100. Higher scores indicate better shoulder function.
Constant-Murley Shoulder Score | 3 weeks after surgery
  The shoulder function was evaluated by the total score of the Constant-Murley Shoulder Score Questionnaire, which ranged from 0 to 100. Higher scores indicate better shoulder function.
Constant-Murley Shoulder Score | 6 weeks after surgery
  The shoulder function was evaluated by the total score of the Constant-Murley Shoulder Score Questionnaire, which ranged from 0 to 100. Higher scores indicate better shoulder function.
Constant-Murley Shoulder Score | 9 weeks after surgery
  The shoulder function was evaluated by the total score of the Constant-Murley Shoulder Score Questionnaire, which ranged from 0 to 100. Higher scores indicate better shoulder function.
Constant-Murley Shoulder Score | 12 weeks after surgery
  The shoulder function was evaluated by the total score of the Constant-Murley Shoulder Score Questionnaire, which ranged from 0 to 100. Higher scores indicate better shoulder function.
Constant-Murley Shoulder Score | 18 weeks after surgery
  The shoulder function was evaluated by the total score of the Constant-Murley Shoulder Score Questionnaire, which ranged from 0 to 100. Higher scores indicate better shoulder function.

SECONDARY OUTCOMES:
Active and passive range of motion | 3 days，1, 2, 3, 6, and 9 weeks after surgery
  In the standard position, the mobility of the shoulder flexion, extension, external rotation and internal rotation was measured by using protractor. The range of flexion is 0-180°, the range of extension is 0-180°, the range of external rotation is 0-90°, and the range of internal rotation is measured. 0-70°. The assessments will be performed in the active and passive state separately.
Shoulder joint muscle strength | 3 days, 3, 6, 9 weeks after surgery
  In the standard position, the muscle strength of the flexion, extension, external rotation and internal rotation of the shoulder joint were assessed according to the "manual muscle test standard".
The power of gripping | 1, 3 days and 1, 2, 3, 6, and 9 weeks after surgery
  In the standard position, the grip of the patient's palm is measured using a dynamometer.
EORTC QLQ BR23 Breast Cancer Quality of Life Questionnaire | 1, 3, 9, 12, 18 weeks after surgery
  The quality of life assessment of breast cancer patients was evaluated by the total score of the EORTC QLQ BR23 Breast Cancer Quality of Life Questionnaire, which ranged from 0 to 92. Higher scores indicate better quality of life.
SF-36 Health status questionnaire | 1, 3, 9, 12, 18 weeks after surgery
  The quality of life assessment of breast cancer patients was evaluated by the total score of the SF-36 Health status questionnaire, which ranged from 0 to 92. Higher scores indicate better quality of life.

OTHER OUTCOMES:
Visual Analogue Scale （VAS) | 1 day, 3 days, 1 week, 2 weeks after surgery
  Visual Analogue Scale（VAS): Used to assess the degree of pain. Draw a 10 cm horizontal line on the paper. One end of the horizontal line is 0, indicating no pain; the other end is 10, indicating severe pain; the middle part indicates different degrees of pain.
Sum drainage from chest wall and axillary after operation. | 1 day, 3 days, 1 week, 2 weeks after surgery
  The postoperative drainage was the total volume of the chest wall drainage tube and the underarm drainage tube. The volume measurement and recording in the drainage bag were observed daily by the nurse.
Upper limb circumference | Preoperative 3, 9, 12,18 weeks after surgery
body weight | Preoperative, 3, 9 weeks after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
The study protocol, statistical analysis plan, informed consent form and clinical study report will be shared online about six months after the trial complete.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: About six months after the trial complete

REFERENCES:
- [Derived] Shu Q, Yang Y, Shao Y, Teng H, Liao R, Li Z, Wu G, Hou J, Tian J. Comparison of Rehabilitation Training at Different Timepoints to Restore Shoulder Function in Patients With Breast Cancer After Lymph Node Dissection: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2023 May;104(5):728-737. doi: 10.1016/j.apmr.2023.01.021. Epub 2023 Feb 20. PMID 36813015
- [Derived] Shao YW, Shu Q, Xu D, Teng H, Wu GS, Hou JX, Tian J. Effect of different rehabilitation training timelines to prevent shoulder dysfunction among postoperative breast cancer patients: study protocol for a randomized controlled trial. Trials. 2021 Jan 6;22(1):16. doi: 10.1186/s13063-020-04954-3. PMID 33407753